CLINICAL TRIAL: NCT01554904
Title: Facial-Flex as a Treatment for Snoring
Brief Title: Study Will Test the Theory That Training With the Facial-Flex Exercise Device Will Improve Snoring in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Facial Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 0102011
Record Dates: First submitted 2012-02-28; First posted 2012-03-15 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Primary Snoring; Sleep Apnea
Keywords: Sleep Study; Snoring; Sleep Apnea; Muscle Laxity; Oral Appliance; Facial Muscles; Neck Muscles; Upper Airway; Muscle Strength; Dynamic Resistance; Oral Exercise; Facial Toning; Facial Muscle Strength; Strap Muscles of the Neck; Apnea-Hypopnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Facial-Flex (Other): The facial flex (FF) exerciser manufactured by Facial Concepts, Inc is an FDA approved Class I medical device for treatment of facial muscle laxity. Facial muscles tend to weaken with age. The combination of deteriorating elastic tissue and facial muscle weakness causes the face to sag. Facial flex consists of two plastic tipped curved lower bars which slide across each other. An external dynamic resistance is provided by elastic bands.
  Interventions: Device: Facial-Flex

INTERVENTIONS:
Device: Facial-Flex — Oral exercise device
  Other Names: Facial Exerciser; Facial Dynamic Resistance; Neck Exerciser

SUMMARY:
The study will test the hypothesis that training with the Facial-Flex exercise device for six weeks will improve snoring in patients with primary snoring or very mild sleep apnea.

DETAILED DESCRIPTION:
Subjects will be studied before and after 6 weeks of Facial-Flex training using portable monitoring. There will be 8 patient visits and 2 additional trips to the sleep center to return the portable sleep monitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of loud snoring but no observed breathing pauses by bed partner (or only very mild obstructive sleep apnea on a previous sleep study within the prior year) will be enrolled.
* Very mild sleep apnea is defined here as an apnea-hypopnea index (AHI) < 10/hour).
* This assumes that the AHI is computed using hypopnea defined as a 30% drop in the flow signal associated with a 4% or greater arterial oxygen desaturation.

Exclusion Criteria:

* Prior upper airway surgery
* Daytime sleepiness (Epworth sleepiness scale >12/24), (obesity BMI > 35 kg/M2)
* Significant arterial oxygen desaturation defined as 5 minutes or more with an arterial oxygen desaturation less than 88%
* Severe insomnia with less than 4 hours of sleep per night
* Uncontrolled psychiatric disorder
* Any disorder causing facial weakness
* Pregnancy
* Temporal mandibular joint problems.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Berry, M.D., Principal Investigator — Professor of Medicine Pulmonary, Critical Care, and Sleep Medicine University of Florida College of Medicine Chief, Pulmonary Section, Malcom Randall VAMC Medical Director, Sleep Disorders Center Shands at AGH
Locations (1):
- Shands Sleep Disorders Center, Gainesville, Florida, United States

REFERENCES:
- [Result] Gary L. Grove, PhD - Skin Study Center, Broomall, PA The Journal of Geriatric Dermatology 1994;2(5):152-158
- [Result] van Lieshout PH, Bose A, Namasivayam AK. Physiological effects of an 8-week mechanically aided resistance facial exercise program. Int J Orofacial Myology. 2002 Nov;28:49-73. PMID 12572260
- [Result] Barry M. Zide, M.D.; James P. Bradley, M.D.;Michael T. Longaker, M.D. Institute of Reconstructive Plastic Surgery at New York University Medical Ctr. Plastic Reconstructive Surgery 2000 March;1154-1158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited at the Shands Sleep Disorders Center through posted advertisement.
Pre-assignment Details: The inclusion and exclusion criteria and study protocol were discussed with potential subjects. Subjects who desired to participate and met criteria signed an informed consent.
Groups:
- Facial-Flex: Subjects meeting inclusion and exclusion criteria who do not have significant obstructive sleep apnea on home sleep study 1 undergo 6 weeks of training with the facial flex (FF) exerciser. At the end of the six weeks of training another sleep study (Home sleep study 2)was performed. The facial flex (FF) exerciser manufactured by Facial Concepts, Inc is an FDA approved Class I medical device for treatment of facial muscle laxity. Facial muscles tend to weaken with age. The combination of deteriorating elastic tissue and facial muscle weakness causes the face to sag. Facial flex consists of two plastic tipped curved lower bars which slide across each other. An external dynamic resistance is provided by elastic bands.
Period: Overall Study
Arm/Group | Facial-Flex
Started | 18
Home Sleep Study 1 | 18 (After informed consent signed.)
Start 6 Weeks of Facial Training | 17 (1 participant was found to have obstructive sleep apnea on the home sleep study #1)
Complete 6 Weeks of Facial Training | 14 (3 subjects withdrew during training)
Home Sleep Study 2 | 14
Completed | 14
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Had sleep apnea on Home Study 1 | 1

BASELINE CHARACTERISTICS:
Population: Number completing study
Arm/Group | Facial-Flex
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 50.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Snore Index
Description: The snore index is the number of snores per hour of monitoring. The pre-treatment and post-treatment (6 weeks) values will be compared. A snore is a vibratory noise usually noted during inspiration and associated with vibration of the uvula and palate. The snore sensor in this study is the nasal pressure cannula connected to a sensitive pressure transducer. Snoring is detected as a fine (high frequency) oscillation superimposed on the nasal pressure waveform. The device [Sleep Scout (ClevMed, Cleveland Ohio)] has an automated scoring detection algorithm to identify breaths with snoring. Each breath with vibration is counted as a snore. As the algorithm is automated and the same snore threshold was used for both baseline and 6 week sleep studies, this prevents technologist bias in detecting snores (breaths with vibration).
Time Frame: baseline and after 6 weeks of facial muscle training
Population: Subjects completing 6 weeks of training and Home Sleep Test # 2
Measure: Mean (Standard Deviation); unit: snores per hour of monitoring
Arm/Group | Facial-Flex
Number analyzed (Participants) | 14
snores per hour of monitoring
  Snore index Sleep study #1 | 348.4 (82.3)
  Snore index Sleep study #2 (after training) | 186.2 (52.2)
Statistical Analysis 1: Comparison: Facial-Flex; The null hypothesis is that the snore index would not be different after 6 weeks of treatment compared to baseline. The comparison group is the subjects completing the 6 weeks of training and the second sleep study; Test type: Superiority or Other; p = 0.02, paired t test; Mean Difference (Final Values) = 162.24, 95% CI 2-sided [27.32 to 297.16], Standard Error of Mean 62.4

2. Secondary Outcome: Apnea-Hypopnea Index (AHI)
Description: The number of apneas and hypopneas per hour of monitoring
Time Frame: baseline and after 6 weeks of facial muscle training
Population: Participants completing 6 weeks of training and second sleep study
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Facial-Flex
Number analyzed (Participants) | 14
events per hour
  Sleep study #1 (baseline) | 3.31 (2.77)
  Sleep study #2 (6 weeks) | 4.16 (4.01)
Statistical Analysis 1: Comparison: Facial-Flex; Participants completing 6 weeks of training and the second sleep study. The null hypothesis was that the AHI would not be different after 6 weeks of training compared to baseline; Test type: Superiority or Other; p = 0.22, t-test, 2 sided — paired t test; Mean Difference (Final Values) = -.85, 95% CI 2-sided [-2.28 to 0.584], Standard Error of Mean 0.66

ADVERSE EVENTS:
Time Frame: Six weeks
Arm/Group | Facial-Flex
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
This was not a sham controlled trial. The number of participants was somewhat limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No